CLINICAL TRIAL: NCT00493376
Title: Prospective Study of Tirapazamine Targeting in Cervical Cancer
Brief Title: Study of Tumour Response to Tirapazamine During Treatment of Cervical Cancer
Status: Terminated | Type: Observational
Why Stopped: This study was a companion study to another one. The other study closed early so this one did as well.
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Other Study IDs: TPZ Targeting Cervix Study
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Cervix Cancer
Keywords: tirapazamine; DNA damage; comet assay
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Glucose Transporter Type 1; Hypoxia-Inducible Factor 1, alpha Subunit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cervical tissue biopsy analysis: Comet assay — Cervical tissue biopsy analysis: Comet assay
Procedure: Biopsy: Measurement of histone gamma H2AX phosphorylation — Biopsy: Measurement of histone gamma H2AX phosphorylation
Procedure: Biopsy: Immunohistochemistry: Ca9, Glut1, HIF-1 alpha — Biopsy: Immunohistochemistry: Ca9, Glut1, HIF-1 alpha
Procedure: Measurement of vascular perfusion: contrast enhanced MRI — contrast enhanced MRI

SUMMARY:
The purpose of this study is as follows:

* to determine whether tirapazamine damages cervical tumour DNA immediately after its administration
* to determine the blood flow and oxygen level of cervical tumour before and after treatment with tirapazamine

DETAILED DESCRIPTION:
Patients with locally advanced cervical cancer can have a poor clinical outcome with standard cisplatin and pelvic radiation therapy. It is well established that pre-treatment tumor hypoxia is a significant prognostic factor in tumors and may be one of the most important and modifiable mechanisms of radiation resistance in this group of tumours. Significant levels of hypoxia are not present in all locally advanced cervical tumors. Hence measurement of the pretreatment tumour oxygenation status is imperative, and can be assessed using various means. Immunohistochemical staining of various intrinsic hypoxia markers to include Ca9, Glut1, HIF-1 alpha on the pre-treatment tumours can be performed.

Tirapazamine, a bio-reductively activated hypoxic cell selective anti-tumour agent, has been found to act synergistically with cisplatinum, resulting in a significantly higher cell kill than expected based on additive action. We proposed to measure the cell killing effect of tirapazamine with the following tests:

* Comet assay: Tirapazamine causes DNA damage that can predict for cell killing by measuring DNA damage in cells from tumor biopsies using the alkaline comet assay.
* Measurement of phosphorylation of histone gamma H2AX: It has been explored as a measure of radiosensitivity in response to clinically relevant doses of radiation. The histone gamma H2AX phosphorylation can be used to detect tirapazamine induced DNA double-strand breaks and collapsed replication forks.

There is some evidence that the drug delivery may be impaired and in fact the drug may not actually be reaching all of the hypoxic tumour cells. A recent study has shown that, in an experimental setting, tirapazamine causes a decrease in vascular perfusion which can be measured with contrast enhanced MRI. We propose to assess if this mechanism is operative in human tumours.

Clinical studies have demonstrated that tumour vascular can increase during the course of radiation therapy, consistent with re-oxygenation and that this is suggestive of a better outcome. Tumours that become less hypoxic during the course of therapy have an increased likelihood of response to the given treatment. However, response to tirapazamine may be reduced. In order to assess both the vascular change that may occur directly because of tirapazamine infusion, as well as any increase in tumour vascularity and perhaps increase in tumour oxygenation during the course of therapy, we plan to assess these tumours during the course of therapy. Assessment of tumour perfusion and vessel permeability after 10 radiation treatments (on day 12) of chemo-radiation therapy will be performed via T1 weighted dynamic contrast enhanced MRI (DCMRI).

We hypothesize that:

1. Tirapazamine (a hypoxic cell cytotoxin and radiosensitizer) will result in increased DNA damage and a better clinical outcome if:

   1. the pre-treatment tumor demonstrates significant hypoxia
   2. tirapazamine treatment results in increased DNA damage
2. tirapazamine acts, in part, by changing vascular perfusion in the tumour and that these changes can be measured with dynamic contrast enhanced MRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed clinically visible invasive carcinoma of the cervix, either squamous cell, adenocarcinoma or a variant of these
* Patients must be enrolled in NCIC CXC.1 (phase 3 study assessing the addition of tirapazamine) and randomized to the tirapazamine arm
* No known bleeding disorder
* Willing to undergo a clinical exam to obtain tissue biopsy for hypoxia marker analysis and DNA damage assessments

Exclusion Criteria:

* Inability to give informed consent
* Criteria below for contrast MRI only :

  1. Chronic renal disease currently on dialysis
  2. Renal insufficiency defined as a Glomerular Filtration Rate (GFR) ≤15cc/min , serum Cr >130, or a BUN>7 measured
  3. Current pacemaker, tens neuro-stimulator, implanted drug infusion devices, any metal implants, foreign metals objects in eyes, aneurysm clips

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Christina Aquino-Parsons, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency, Vancouver Centre, Vancouver, British Columbia, Canada